CLINICAL TRIAL: NCT02867488
Title: Dose-response Effects of Soybean Oil in Salad Dressing on Carotenoid/Fat-soluble Vitamin Bioavailability in Salad Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Wendy S. White, Associate Professor, Iowa State University
Other Study IDs: 08-549
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Biological Availability
Keywords: carotenoids; phylloquinone; tocopherols; vitamin A
MeSH Terms: interventions — Soybean Oil; Condiments

INTERVENTIONS:
Other: Soybean oil in salad dressing

SUMMARY:
The objectives will be to evaluate the dose-response between the amount of soybean oil in salad dressing and the absorption of: 1) carotenoids, phylloquinone, and tocopherols in salad vegetables; 2) retinyl palmitate formed from the provitamin A carotenoids, alpha- and beta-carotene.

ELIGIBILITY:
Inclusion Criteria:

* General good health as determined by interview, blood biochemistry profile, complete blood count, and plasma lipid and lipoprotein profile

Exclusion Criteria:

* Cigarette smoking, frequent alcohol consumption
* Use of vitamin/mineral supplements
* Lactose intolerance
* Known food allergies
* Body mass index (BMI) 30 or higher
* Eating disorder or restrained eating
* Vegetarianism
* Hyperlipidemia
* Current or planned pregnancy
* Use of hormonal contraceptives (affects chylomicron clearance); use of plant sterols or medications known to affect lipid metabolism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve for carotenoids, phylloquinone, tocopherols, and retinyl palmitate in the plasma chylomicron fraction | 0-9.5 hours postprandially

REFERENCES:
- [Derived] White WS, Zhou Y, Crane A, Dixon P, Quadt F, Flendrig LM. Modeling the dose effects of soybean oil in salad dressing on carotenoid and fat-soluble vitamin bioavailability in salad vegetables. Am J Clin Nutr. 2017 Oct;106(4):1041-1051. doi: 10.3945/ajcn.117.153635. Epub 2017 Aug 16. PMID 28814399